CLINICAL TRIAL: NCT01398293
Title: A Single-center, Single-dose, Randomized, Double-blind, Double-dummy, Placebo-controlled, Positive-controlled, Four-way Crossover Study to Investigate the Effect of Danoprevir With Low Dose Ritonavir (DNV/r) on the QT/QTc Interval in Healthy Subjects
Brief Title: A Study of Danoprevir in Combination With Low-Dose Ritonavir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: NP25298; 2011-001413-13 (EudraCT Number)
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Moxifloxacin; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Experimental)
  Interventions: Drug: danoprevir; Drug: moxifloxacin placebo; Drug: ritonavir
- B (Experimental)
  Interventions: Drug: danoprevir; Drug: moxifloxacin placebo; Drug: ritonavir
- C (Active Comparator)
  Interventions: Drug: danoprevir placebo; Drug: moxifloxacin; Drug: ritonavir placebo
- D (Placebo Comparator)
  Interventions: Drug: danoprevir placebo; Drug: moxifloxacin placebo; Drug: ritonavir placebo

INTERVENTIONS:
Drug: danoprevir — 100 mg single dose orally
  Arms: A
Drug: danoprevir — 400 mg single dose orally
  Arms: B
Drug: danoprevir placebo — single oral dose
  Arms: C; D
Drug: moxifloxacin — 400 mg single dose orally
  Arms: C
Drug: moxifloxacin placebo — single oral dose
  Arms: A; B; D
Drug: ritonavir — 100 mg single dose orally
  Arms: A; B
Drug: ritonavir placebo — single oral dose
  Arms: C; D

SUMMARY:
This single-dose, randomized, double-blind, double-dummy, placebo-controlled, positive-controlled four-way crossover study will evaluate the effect of a single dose of danoprevir with low-dose ritonavir on the QC/QTc interval in healthy volunteers. Subjects will be randomly assigned to one of four sequences with treatments of A: therapeutic dose of danoprevir plus ritonavir (DNV/r), B: supratherapeutic dose of DNV/r, C: moxifloxacin and D: placebo, with a washout period of at least 7 days between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers, 18 - 60 years of age
* Female subjects must be surgically sterile or post-menopausal
* Male subjects and their partners of child-bearing potential must use to methods of contraception for the duration of the study and for three months after the last drug administration
* Agree to abstain from strenuous exercise for three days before dosing and throughout the study (including washout period and follow-up visit)

Exclusion Criteria:

* History or evidence of any clinically significant disease or disorder
* Pregnant or lactating women
* Male partners of women who are lactating or trying to become pregnant
* Current smokers or subjects who have discontinued smoking less than six months prior to first dosing
* Positive alcohol breath test; suspicion of regular consumption of drugs of abuse
* Positive for hepatitis B, hepatitis C or HIV infection
* Participation in an investigational drug, biologic, or device study within three months before first study drug administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Threshold pharmacological effect on cardiac repolarization as detected by changes in the QT/QTc interval following single dose | approximately 9 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Plasma concentrations | approximately 9 weeks
Safety: Incidence of adverse events | approximately 9 weeks
Cardiac response: Electrocardiogram (ECG) | approximately 9 weeks
Correlation between pharmacokinetics (plasma concentrations) and QT/QTc interval changes | approximately 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Strasbourg, France